CLINICAL TRIAL: NCT01864434
Title: In Vivo Comparison of Kinematics for Patients Implanted With Either a Stryker or a Zimmer Posterior Cruciate Retaining Total Knee Arthroplasty
Brief Title: In Vivo Kinematics Comparison of Stryker or Zimmer Total Knee Arthroplasty
Status: Completed | Type: Observational
Sponsor: The University of Tennessee, Knoxville (Other)
Collaborators: Stryker Orthopaedics (Industry)
Responsible Party: Principal Investigator, Richard Komistek, Principal Investigator, The University of Tennessee, Knoxville
Other Study IDs: 130180/2012017; R011373454 (Other Grant/Funding Number: Stryker Orthopaedic)
Record Dates: First submitted 2013-05-16; First posted 2013-05-29 (Estimated); Results first posted 2014-12-24 (Estimated); Last update posted 2019-10-10 (Actual); Status verified 2019-10

CONDITIONS: Knee Prosthesis
Keywords: Knee Prosthesis; Total Knee Arthroplasty; Cruciate Retaining; Posterior Cruciate Retaining
MeSH Terms: interventions — Polymerase Chain Reaction; Arthroplasty, Replacement, Knee

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with a Stryker Triathlon CR TKA: Patients implanted with a Stryker Triathlon Posterior Cruciate Retaining Total Knee Arthroplasty.
  Interventions: Device: Stryker posterior cruciat retaining (PCR) total knee arthroplasty (TKA)
- Patients with a Zimmer PCR TKA: Patients implanted with a Zimmer NexGen Posterior Cruciate Retaining Total Knee Arthroplasty.
  Interventions: Device: Zimmer PCR TKA

INTERVENTIONS:
Device: Stryker posterior cruciat retaining (PCR) total knee arthroplasty (TKA) — The fluoroscopy procedure itself is used as a means of data collection and is not the intervention under investigation; therefore, the study is observational and not interventional.
  Other Names: Triathlon PCR TKA
  Groups: Patients with a Stryker Triathlon CR TKA
Device: Zimmer PCR TKA — The fluoroscopy procedure itself is used as a means of data collection and is not the intervention under investigation; therefore, the study is observational and not interventional.
  Other Names: Zimmer NexGen PCR TKA
  Groups: Patients with a Zimmer PCR TKA

SUMMARY:
This study will compare the kinematics data collected from patients with implants created by different manufacturers to see which of these implants provides a more normal-like kinematic pattern compared to the normal knee.

DETAILED DESCRIPTION:
A better understanding of knee joint kinematics is important to explain premature polyethylene wear failures within knee implants and to help design a prosthesis that most closely approximates the normal knee. Therefore, the objectives for this study are to compare the in vivo kinematic patterns for subjects implanted with either a Stryker Triathlon Posterior Cruciate Retaining (PCR) Total Knee Arthroplasty (TKA) or Zimmer NexGen PCR TKA design to determine if there are any kinematic differences between these TKA designs. Each subject will be asked to undergo a fluoroscopic evaluation while performing weight-bearing activities under surveillance using the University of Tennessee's new mobile tracking fluoroscopic unit while performing deep knee bend and ramp up and ramp down activities. The mobile fluoroscopy unit is approved for use by the State of Tennessee on a study-by-study basis after IRB approval is obtained for each study.

ELIGIBILITY:
Inclusion Criteria:

* Must be at least 3 months post-operative with no other surgical procedures conducted within the past 6 months
* Must have body weight of less than 250 lbs
* Must have Body Mass Index of less than 38
* Must be judged clinically successful with a Knee Society Score >90
* Must have 100% post-operative passive flexion with no ligamentous laxity or pain
* Must be able to walk on level ground without aid of any kind
* Must be able to ascend and descend a ramp with a 10 degree incline with no assistance
* Must be willing to sign both Informed Consent and HIPAA forms
* Must be between 160 cm (5'3) and 193 cm (6'4) tall

Exclusion Criteria:

* Pregnant or potentially pregnant females
* Unwilling to sign Informed Consent or HIPAA forms

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be patients of Dr. Harold E. Cates of Tennessee Orthopaedic Clinics and must have been implanted with either a Stryker Triathlon CR TKA or Zimmer PCR TKA
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2013-06; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adrija Sharma, Ph D, Principal Investigator — The University of Tennessee; Richard D Komistek, Ph D, Principal Investigator — The University of Tennessee; William R Hamel, Ph D, Principal Investigator — The University of Tennessee; Harold E Cates, MD, Principal Investigator — Tennessee Orthopaedic Clinics
Locations (4):
- United States (4):
  - Tennessee Orthopaedic Clinic, Tennessee Orthopaedic Foundation for Education & Research, Knoxville, Tennessee
  - Dougherty Engineering Building, Room M007, Knoxville, Tennessee
  - Perkins Hall, The University of Tennessee, Knoxville, Tennessee
  - Science and Engineering Research Facility, Knoxville, Tennessee

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients With a Stryker Triathlon CR TKA: Patients implanted with a Stryker Triathlon Cruciate Retaining Total Knee Arthroplasty.
  Stryker PCR TKA
- Patients With a Zimmer PCR TKA: Patients implanted with a Zimmer Poster Cruciate Retaining Total Knee Arthroplasty.
  Zimmer PCR TKA
Period: Overall Study
Arm/Group | Patients With a Stryker Triathlon CR TKA | Patients With a Zimmer PCR TKA
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Patients With a Stryker Triathlon CR TKA | Patients With a Zimmer PCR TKA | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 7 | 14
  >=65 years | 18 | 18 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.7 (6.4) | 70.6 (9.4) | 69.60 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 19 | 21
  Male | 23 | 6 | 29
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Kinematics - Deep Knee Bend Activity
Description: Lateral Anterior Posterior (LAP) and Medial Anterior Posterior (MAP) translations, and Axial Rotation (AR) and maximum flexion of medial femoral condyles during deep knee bend (DKB) activity
Time Frame: 3 months post-operative
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Patients With a Stryker Triathlon CR TKA | Patients With a Zimmer PCR TKA
Number analyzed (Participants) | 25 | 25
mm
  Lateral Anterior Posterior Deep Knee Bend | -0.43 (3.43) | -1.00 (3.23)
  Medial Anterior Posterior Deep Knee Bend | 3.51 (2.68) | -0.42 (2.20)
  Axial Rotation Deep Knee Bend | 5.20 (3.93) | 0.75 (5.12)
  Maximum Flexion Deep knee bend | 107.80 (8.50) | 107.20 (11)

2. Primary Outcome: Kinematics - Ramp up Activity
Description: Lateral Anterior Posterior (LAP) [during 3 moments - 0-33%, 33-66% and 66-100%] and Medial Anterior Posterior (MAP) [during 3 moments - 0-33%, 33-66% and 66-100%] translations, and Axial Rotation (AR) [during 3 moments - 0-33%, 33-66% and 66-100%] of medial femoral condyles during ramp up activity
Time Frame: 3 months post-operative
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Patients With a Stryker Triathlon CR TKA | Patients With a Zimmer PCR TKA
Number analyzed (Participants) | 25 | 25
mm
  Lateral Anterior Posterior Translation 0% to 33% | -0.31 (2.41) | 0.20 (2.75)
  Lateral Anterior Posterior Translation 33% to 66% | -0.94 (2.26) | -0.61 (2.42)
  Lateral Anterior Posterior Translation 66% to 100% | -0.23 (2.69) | -0.07 (2.70)
  Medial Anterior Posterior Translation 0% to 33% | -1.31 (3.43) | -1.88 (2.07)
  Medial Anterior Posterior Translation 33% to 66% | -1.04 (3.36) | 0.41 (2.16)
  Medial Anterior Posterior Translation 66% to 100% | 0.48 (2.35) | -0.09 (1.63)
  Axial Rotation 0% to 33% | -1.33 (4.03) | -2.69 (3.99)
  Axial Rotation 33% to 66% | -0.15 (3.17) | 1.27 (3.42)
  Axial Rotation 66% to 100% | 0.95 (2.19) | -0.03 (3.96)

3. Primary Outcome: Kinematics - Ramp Down Activity
Description: Lateral Anterior Posterior (LAP) [during 3 moments - 0-33%, 33-66% and 66-100%] and Medial Anterior Posterior (MAP) [during 3 moments - 0-33%, 33-66% and 66-100%] translations, and Axial Rotation (AR) [during 3 moments - 0-33%, 33-66% and 66-100%] of medial femoral condyles during ramp down activity
Time Frame: 3 months post-operative
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Patients With a Stryker Triathlon CR TKA | Patients With a Zimmer PCR TKA
Number analyzed (Participants) | 25 | 25
mm
  Lateral Anterior Posterior Translation 0% to 33% | -0.57 (2.33) | -1.11 (2.27)
  Lateral Anterior Posterior Translation 33% to 66% | -1.25 (1.86) | -0.96 (2.6)
  Lateral Anterior Posterior Translation 66% to 100% | 0.83 (2.56) | 0.15 (2.37)
  Medial Anterior Posterior Translation 0% to 33% | -0.87 (2.19) | -0.92 (1.95)
  Medial Anterior Posterior Translation 33% to 66% | -.75 (2.42) | 0 (1.27)
  Medial Anterior Posterior Translation 66% to 100% | 1.29 (2.34) | -0.31 (1.44)
  Axial Rotation 0% to 33% | -0.44 (2.76) | 0.24 (3.19)
  Axial Rotation 33% to 66% | 0.67 (3.09) | 1.22 (3.97)
  Axial Rotation 66% to 100% | 0.59 (3.39) | -0.54 (3.86)

ADVERSE EVENTS:
Arm/Group | Patients With a Stryker Triathlon CR TKA | Patients With a Zimmer PCR TKA
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes